CLINICAL TRIAL: NCT05395936
Title: Mastectomy Flap Temperature and Clinical Implications
Brief Title: Mastectomy Flap Temperature Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00075787; WFBCCC 74222 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Data Collection Arm (Experimental): Participants scheduled for mastectomy with or without breast reconstruction during the course of their breast surgery treatment will have breast skin temperatures taken using a myocardial probe in different anatomical breast areas at multiple time points during the surgery.
  Interventions: Other: Myocardial Probe Temperature Screen; Other: Data Collection

INTERVENTIONS:
Other: Myocardial Probe Temperature Screen — The myocardial probe is a needle that measures temperatures. The skin site for introducing the myocardial probe will be small enough that participants will not notice that temperatures have been collected. If participants have multiple operations, temperatures may be collected at each operation.
Other: Data Collection — Study team members will collect medical history and other information to potentially understand the safety and success of breast surgery better to allow investigators to identify variables, or changes to help understand investigators roles in potential complications in breast surgery.

SUMMARY:
The purpose of this research study is to measure tissue temperatures and generate a prospective database of participants undergoing mastectomy with or without breast reconstruction at Wake Forest Baptist Hospital (WFBH) in order to enable and facilitate the evaluation of important and novel research questions - and quality improvement (QI) ideas/objectives - that may improve the care of breast surgery patients.

DETAILED DESCRIPTION:
Primary Objective(s)

* Quantify the proportion of eligible women approached who consent to intraoperative (pre and post mastectomy) measurement of mastectomy flap temperatures in each of 4 quadrants of each relevant breast (i.e., unilateral or bilateral procedure).
* Quantify the proportion of patients upon whom the surgical team is able to obtain intraoperative flap measurements from each of 4 quadrants on each relevant breast pre- and post-mastectomy and pre-implant.

Secondary Objective: To measure mastectomy flap temperatures in 4 quadrants pre-mastectomy, following mastectomy, and pre-implant, and compare average flap temperature to average core body temperature.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral or bilateral mastectomy with implant based breast reconstruction within the Wake Forest Baptist Health System.
* Aged 18 or older.
* Ability to understand an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria: Those who are male.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Katz, MD, Principal Investigator — Wake Forest Baptist Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Data Collection Arm
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Data Collection Arm
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Consenting to Have Mastectomy Flap Temperatures Measured During Surgery
Description: This will be computed by the dividing the total number of eligible women screened by the number of women who consent.
Time Frame: 90 days post surgery
Population: 22 eligible women were approached to participate, 19 agreed to participate in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Data Collection Arm
Number analyzed (Participants) | 22
Participants | 19

2. Primary Outcome: Number of Women Having All Relevant Flap Temperatures Measured
Description: This will either be 12 or 24 total expected flap temperatures: 4 quadrants, at three time points- pre and post-mastectomy and pre-implant placement; one or both breasts), and we will compute a 95% confidence interval.
Time Frame: 90 days post surgery
Population: Temperature measurements were only obtained for 15 of the participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Data Collection Arm
Number analyzed (Participants) | 19
Participants | 15

3. Secondary Outcome: Change in Mastectomy Flap Temperatures and Core Body Temperatures
Description: Mastectomy flap temperatures will be measured using a 22 gauge myocardial temperature sensor (Smiths Medical). Temperatures will be recorded in degrees Celsius. Core body temperature will also be collected to observe a difference between pre and post-mastectomy average mean flap temperature, average core body temperature and pre-implant average core body temperature and flap temperature readings.
Time Frame: At pre-mastectomy (baseline), pre-implant (before surgery) and post mastectomy (up to 90 days post surgery)
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Intraoperative Data Collection Arm
Number analyzed (Participants) | 19
Degrees Celsius
  Pre-mastectomy average core temperature readings | 35.3 (1.6)
  Pre-mastectomy average flap temperature readings | 30.4 (1.7)
  Post-mastectomy average core temperature readings | 35.6 (1.7)
  Post-mastectomy average flap temperature readings | 29.9 (2.0)
  Pre-implant average core body temperature readings | 35.9 (0.5)
  Pre-implant average flap temperature readings | 29.0 (1.9)
Statistical Analysis 1: Comparison: Intraoperative Data Collection Arm; Test type: Superiority; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants will be followed for 90 days after surgery for adverse events
Arm/Group | Intraoperative Data Collection Arm
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT05395936/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT05395936/ICF_000.pdf